CLINICAL TRIAL: NCT00920946
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Safety and Efficacy Study of Dimebon in Patients With Mile-to-Moderate Huntington Disease
Brief Title: A Safety and Efficacy Study of Dimebon in Patients With Huntington Disease
Acronym: HORIZON
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medivation, Inc. (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DIM20
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Huntington Disease
Keywords: Huntington; Dimebon; HD; Huntingtin
MeSH Terms: conditions — Huntington Disease | interventions — latrepirdine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- Dimebon (Experimental)
  Interventions: Drug: Dimebon

INTERVENTIONS:
Drug: Dimebon — 20 mg Dimebon orally TID
  Arms: Dimebon
Other: Placebo — Orally TID
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if Dimebon is safe and effective for the treatment of cognitive impairment in Huntington disease.

DETAILED DESCRIPTION:
This study is a multicenter Phase 3, randomized, double-blind, placebo-controlled safety and efficacy study of Dimebon treatment in subjects with Huntington disease (HD). The study will evaluate Dimebon 20 mg three times daily (TID) administered orally (PO) for six months (26 weeks) compared with matching placebo TID for the primary safety and efficacy analyses. Safety and tolerability will be assessed by recording of adverse events and by monitoring of vital signs, physical examinations, safety laboratory evaluations, and 12-lead electrocardiogram(ECG)assessments.

ELIGIBILITY:
Inclusion Criteria:

* Have clinical features of HD and a CAG polyglutamate repeat expansion ≥ 36
* Have cognitive impairment as noted by the following:

  1. A Screening MMSE AND a baseline (pre-dose) MMSE score between 10 and 26 (inclusive); and
  2. A subjective assessment of cognitive impairment with decline from pre-HD levels by the Investigator after interviewing the subject and caregiver;
* Are willing and able to give informed consent
* Aged 30 years or older
* Have a caregiver who assists/spends time with the subject at least five days per week for at least three hours per day and has intimate knowledge of the subject's cognitive, functional, and emotional states, and of the subject's personal care.

Exclusion Criteria:

* Had onset of symptoms prior to age 18
* Have any major medical illness or unstable medical condition within 180 days of screening that may interfere with the subject's ability to comply with study procedures and abide by study restrictions, or with the ability to interpret safety data

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2009-07; Primary Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
A comparison between the mean changes from baseline in the Dimebon 20 mg TID treatment group and the placebo group on the MMSE | Week 26
A comparison of the distributions of the CIBIC-plus (ADCS CGIC)in the Dimebon 20 mg TID treatment group and the placebo group | Week 26

SECONDARY OUTCOMES:
A comparison between the mean changes from baseline of the Dimebon 20 mg TID treatment group and the placebo group on the NPI | Week 26
A comparison between the mean changes from baseline of the Dimebon 20 mg TID treatment group and the placebo group on the ADCS-ADL | Week 26
A comparison between the mean changes from baseline of the Dimebon 20 mg TID treatment group and the placebo group on the UHDRS'99 Total Motor Score | Week 26

CONTACTS AND LOCATIONS:
Locations (37):
- United States (24):
  - Scottsdale, Arizona
  - Davis, California
  - Irvine, California
  - La Jolla, California
  - San Francisco, California
  - Gainsville, Florida
  - Miami, Florida
  - Boise, Idaho
  - Indianapolis, Indiana
  - Kansas City, Kansas
  - Wichita, Kansas
  - Charlestown, Massachusetts
  - Golden Valley, Minnesota
  - St Louis, Missouri
  - New York, New York
  - Rochester, New York
  - Durham, North Carolina
  - Winstom-Salem, North Carolina
  - Cleveland, Ohio
  - Columbus, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Milwaukee, Wisconsin
- Australia (3):
  - Wentworthville, New South Wales
  - Melbourne, Victoria
  - Perth
- Canada (3):
  - Vancouver, British Columbia
  - London, Ontario
  - Montreal, Quebec
- Copenhagen, Denmark
- Germany (4):
  - Oberer Eslebberg, Ulm
  - Aachen
  - Bochum
  - Hamburg
- Stockholm, Sweden
- Birmingham, United Kingdom

REFERENCES:
- [Derived] HORIZON Investigators of the Huntington Study Group and European Huntington's Disease Network. A randomized, double-blind, placebo-controlled study of latrepirdine in patients with mild to moderate Huntington disease. JAMA Neurol. 2013 Jan;70(1):25-33. doi: 10.1001/2013.jamaneurol.382. PMID 23108692
- See also: Study website — http://www.horizontrial.com